CLINICAL TRIAL: NCT02146820
Title: LASER TREATMENT OF BENIGN PIGMENTED LESIONS WITH A DUAL WAVELENGTH PICOSECOND LASER
Brief Title: Picosecond Laser for Ttreatment of Benign Pigmented Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DHF13661
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Benign Pigmented Lesions
Keywords: Pigmented Lesions, Skin Pigment, Picosecond Laser, Syneron
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Picosecond Laser System (Experimental)
  Interventions: Device: GentleMax system

INTERVENTIONS:
Device: GentleMax system — Picosecond Laser System for the Treatment of Pigmented Lesions

SUMMARY:
The purpose of this study is to determine whether Pico laser is effective and safe in the treatment of benign pigmented lesions.

DETAILED DESCRIPTION:
The Investigational device is a dual wavelength laser system developed for treatment of pigmented lesions and for tattoo removal. The base unit is a GentleMax system modified to emit light at wavelengths of 532 and 1064 nm and deliver pulse energy up to 400mJ, and pulse duration of 700 ps.

ELIGIBILITY:
Inclusion Criteria:

1. Has Fitzpatrick skin type I-VI
2. Has unwanted benign pigmented lesions including but not limited to solar lentigines, freckles, café au lait, melasma, New of Ota, Nevus of Ito, and hyperpigmentation, and wishes to undergo laser treatments to remove them
3. Is willing to sign an informed consent form to participate in the study
4. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits

Exclusion Criteria:

1. Is hypersensitive to light exposure
2. Has an active sun tan
3. Has active localized or systemic infection
4. Is taking medication(s) for which sunlight is a contraindication
5. Has a history of squamous cell carcinoma or melanoma
6. Has a history of keloid scarring
7. Has used oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment, e.g., lack of noticeable skin flaking, skin peeling and skin surface roughness.
8. Has had a laser procedure, a peel or has used lightening creams in the area to be treated with in the past six months
9. Has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications
10. Is female and pregnant is currently breast feeding or planning a pregnancy during the study period
11. Is allergic to lidocaine, tetracaine or Xylocaine with epinephrine
12. Subjects with pigmented lesions that are considered not acceptable by the study doctor or any condition that, in the study doctor's opinion, would make it unsafe to treat.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Global percentage of pigment clearance | 3 months post the final treatment
  Global percentage of pigment clearance evaluated by blinded observers using post treatment photographs compared to baseline photographs.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 3 months
  Adverse events will be evaluated immediately after and before each subsequent laser treatment and will be based on the incidence and severity of side effects caused by the laser treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Mann, Study Director — Syneron Medical Ltd.
Locations (2):
- Laser and Cosmetic Dermatology, San Francisco, California, United States
- Hong Kong Dermatology and Laser Centre, Hong Kong, China